CLINICAL TRIAL: NCT00113022
Title: An Investigation of the Antidepressant Efficacy and Safety of an AMPAkine (Org 24448) in Major Depressive Disorder, A Double-Blind, Placebo-Controlled, Randomized Study
Brief Title: Org 24448 to Treat Major Depression
Status: Terminated | Phase: Phase 2 | Type: Interventional
Why Stopped: Terminated due to concerns about adverse events in separate study.
Sponsor: National Institute of Mental Health (NIMH) (NIH)
Responsible Party: Carlos A. Zarate, M.D./National Institute of Mental Health, National Institutes of Health
Organization: National Institutes of Health Clinical Center (CC) (NIH)
Allocation: Randomized | Model: Parallel | Masking: Quadruple | Purpose: Treatment
Other Study IDs: 050161; 05-M-0161 (Other: CNS-IRB, NIH)
Record Dates: First submitted 2005-06-02; First posted 2005-06-03 (Estimated); Results first posted 2012-07-06 (Estimated); Last update posted 2012-07-13 (Estimated); Status verified 2012-07

CONDITIONS: Depression
Keywords: Depression; Glutamate; Ampakine; Treatment; Memory; Major Depressive Disorder; AMPA Receptor Activation; BDNF
MeSH Terms: conditions — Depression; Depressive Disorder, Major | interventions — 1-(benzofurazan-5-ylcarbonyl)piperidine

STUDY DESIGN:
Who Masked: Participant, Care Provider, Investigator, Outcomes Assessor
Oversight: Data Monitoring Committee: Yes

ARMS (2):
- Org 24448 (Experimental): Blinded, active experimental compound
  Interventions: Drug: Org 24448
- Placebo (Placebo Comparator): Blinded placebo
  Interventions: Drug: Placebo

INTERVENTIONS:
Drug: Org 24448 — 250 mg once per day for first week, 250 mg twice per day for second week, 500 mg twice per day for third and fourth weeks, if response minimal or worse at four weeks then 750 mg twice per day for additional weeks
  Other Names: Ampakine
  Arms: Org 24448
Drug: Placebo — Inactive equivalent of 250 mg once per day for first week, 250 mg twice per day for second week, 500 mg twice per day for third and fourth weeks, if response minimal or worse at four weeks then 750 mg twice per day for additional weeks
  Arms: Placebo

SUMMARY:
This study will evaluate the effectiveness of the experimental drug, Org 24448, for short-term treatment of depression. It will examine the effects of the drug on symptoms, such as low mood and persistent sadness, poor sleep and appetite, poor motivation and lack of enjoyment of things people normally enjoy, negative thinking, and feeling slowed down or having trouble concentrating. It will also assess whether the drug improves cognitive function, especially memory.

Patient with major depression who do not have a serious, unstable medical illness and who are 21 to 55 years of age may be eligible for this study. Candidates are screened with a psychiatric and medical history, diagnostic interview, physical examination, electrocardiogram, blood tests and, for women, a pregnancy test.

Participants are tapered off anti-depression drugs (and any other medications not allowed on the study) over a 3-week period and then begin a 2-week drug-free period. During these 2 weeks they have an electroencephalogram (EEG) with light stimulation, and those whose EEG indicates a seizure disorder are excluded from the study. Also at the beginning of the drug-free period they begin taking a placebo ("sugar pill") twice a day. After 2 weeks on placebo, some patients begin treatment with Org 24448, while others remain on placebo. They continue the medication for 8 weeks, during which time they have a weekly check of vital signs, blood and urine tests, and rating scales for depression and anxiety. Level of functioning is evaluated twice during the study. After 8 weeks of treatment, patients have a physical exam, electrocardiogram (ECG), EEG, blood tests, and begin to come off the study drug, tapering the medication over a week.

In addition to the above procedures, some patients undergo the following tests during the 2-week drug-free period and again toward the end of the 8-week medication phase:

* Neuropsychological testing, including measurements of cognitive abilities such as memory, attention, problem-solving, and language skills.
* Positron emission tomography (PET): This nuclear medicine test provides information about different brain regions. The patient lies on a table in the PET scanner (similar to a computed tomography (CT) scanner), with a mask placed over his or her face that helps keep the head still. A sugar fluid with a radioactive material attached to it is injected into a catheter (plastic tube) that has been inserted into a vein in the patient's arm. The scanner detects ...

DETAILED DESCRIPTION:
Depression is a devastating illness that is estimated to affect 12% to 17% of the population at some point during the lifetime of an individual. Despite the availability of a wide range of antidepressant drugs, 30% to 40% of patients with major depression fail to respond to first-line antidepressant (e.g., selective serotonin reuptake inhibitors (SSRIs)) treatment, despite adequate dosage, duration, and compliance. Thus there is a clear need to develop novel and improved therapeutics for major depression. Current pathophysiological theories regarding the neurobiology of depression include alterations in intracellular signaling cascades, and impairments of cellular plasticity and resilience. There is recent evidence suggesting that promoting growth factors such as brain derived neurotrophic factor (BDNF) may provide a mechanism for the treatment of depression. New information indicating modulation of glutamate receptors in the actions of antidepressant treatments suggests a novel approach to develop a new class of antidepressants. Studies have shown that the biarylpropylsulfonamide AMPA (2-amino-3-(5-methyl-3-oxo-1,2-oxazol-4-yl) propanoic acid) receptor potentiators (LY392098 and LY451616) have antidepressant effects in animal models of depression. Several studies have demonstrated that AMPA receptor activation can increase expression of BDNF both in vitro and in vivo. Thus, one possible new approach for the treatment of depression is to use an AMPA receptor potentiator.

In this study we propose to compare the ampakine receptor potentiator Org 24448 to placebo for the treatment of Major Depression. Inpatients and outpatients (primarily outpatients), ages 21 to 70, with a diagnosis of Major Depression (without psychotic features), will be randomized to double-blind treatment to either Org 24448 or placebo for a period of 8 weeks. Acute efficacy will be determined by demonstrating a greater response rate using specified criteria. Approximately 90 patients with acute major depression will be enrolled in the study in order to reach the goal of randomizing 70 patients in the controlled trial.

ELIGIBILITY:
INCLUSION CRITERIA:

1. Male or female subjects, 21 to 70 years of age.
2. Female subjects who are not of childbearing potential (i.e., surgically sterile, postmenopausal for at least one year) or must be using a medically accepted means of contraception. Women using oral contraceptive medication for birth control must also be using a barrier contraceptive. Women of childbearing potential must also have a negative serum Beta-HCG (human chorionic gonadotropin) at pre-study.
3. Subjects must fulfill DSM-IV criteria for Major Depression (296.3) without psychotic features, based on clinical assessment and confirmed by a structured diagnostic interview, the Structured Clinical Interview for DSM-IV TR Axis I Disorders, SCID-P.
4. Subjects have a history of at least one previous episode of depression prior to the current episode.
5. Subjects must have an initial score of greater than or equal to 32 on the Inventory of Depressive Symptoms, Clinician version (IDS-C) at Visit 1 and Visit 2.
6. Subjects must not have greater than a 25% decrease in the IDS-C total scores during washout (between Visits 1 and 2).
7. Each subject must have a level of understanding sufficient to agree to all tests and examinations required by the protocol and must sign an informed consent document.
8. Current major depressive episode of at least 4 weeks duration.
9. Subjects who have not responded to adequate previous trials of at least one antidepressant as determined by the Antidepressant Treatment History Form (ATHF) criteria (score greater than or equal to 3). Additionally, patients who have not completed antidepressants trials of adequate dose and duration due to intolerance to therapy may be induced if they have demonstrated intolerance to greater than or equal to 3 antidepressant medications in the current or a previous episode, and did not meet ATHF criteria for a single adequate treatment trial in the current episode. 3 intolerant trials would count as an adequate failed trial. If this criteria has not been met, the Principal Investigator may allow for a four-week prospective trial of a standard antidepressant (at the patients' and clinicians' discretion) for potential participants who have not responded to at least one adequate trial for the current episode per inclusion criteria.

   EXCLUSION CRITERIA:
10. Presence of psychotic features or a diagnosis of Schizophrenia or any other psychotic disorder or bipolar disorder as defined in the Diagnostic and Statistical Manual, Version IV (DSM-IV).
11. Subjects with a diagnosis of Obsessive Compulsive Disorder as defined in the DSM-IV.
12. Subjects reporting Borderline or Antisocial Personality disorders. Other Axis II disorders do not qualify one for exclusion from the study.
13. Subjects with a history of DSM-IV drug or alcohol dependency or abuse (except for nicotine or caffeine) within the preceding 3 months.
14. Female subjects who are either pregnant or nursing.
15. Serious, unstable illnesses including hepatic, renal, gastroenterologic, respiratory, cardiovascular (including ischemic heart disease), endocrinologic, neurologic, immunologic, or hematologic disease.
16. Subjects with a history of neutropenia or medication-induced blood dyscrasia.
17. Clinically significant abnormal findings of laboratory parameters, physical examination, EEG, or ECG.
18. Subjects with a lifetime history of autism, mental retardation, pervasive developmental disorders, or Tourette's syndrome.
19. Subjects with uncorrected hypothyroidism or hyperthyroidism.
20. Subjects with one or more seizures without a clear and resolved etiology.
21. Treatment with a reversible monoamine oxidase inhibitor (MAOI) within 2 weeks prior to Visit 2.
22. Treatment with fluoxetine within 4 weeks prior to Visit 2.
23. Treatment with clozapine or electroconvulsive therapy (ECT) within 3 months prior to study Visit 2.
24. Judged clinically to be at serious suicidal or homicidal risk.
25. Participation in a clinical trial of another investigational drug within 1 month prior to study entry (visit 1).
26. Patients starting hormonal treatment (e.g., estrogen) in the last 3 months prior to visit 1.
27. Patients undergoing current nonpharmacologic antidepressant treatments, such as light therapy and psychotherapy.
28. Patients will be excluded who have previously failed greater than or equal to 3 lifetime adequate antidepressant trials by ATHF criteria (Sackeim 2001).
29. Patients with any evidence of a seizure disorder as assessed by an EEG with photic stimulation.

ADDITIONAL INCLUSION AND EXCLUSION CRITERIA FOR PET SCANS ONLY: THIRTY SUBJECTS WITH MAJOR DEPRESSIVE DISORDER WILL PARTICIPATE IN THE IMAGING COMPONENT OF THIS STUDY.

INCLUSION:

1. Subjects who are ages 21-70.
2. Subjects with an early age of onset (before age 40).
3. Subjects who either meet melancholic subtype criteria and/or have a first degree relative with bipolar disorder.
4. Negative pregnancy test within 24 hours of positron emission tomography (PET) in women of childbearing potential.

EXCLUSION:

1. Subjects will have been off psychotropic drugs (including zolpidem) for at least 3 weeks (8 weeks for fluoxetine) prior to PET.
2. Subjects with a history of lifetime DSM-IV substance dependence (except for nicotine or caffeine).
3. Subjects with substance abuse within 12 months (except for nicotine or caffeine).
4. Subjects with a current or lifetime history of hypertension or diabetes.
5. Subjects who have reached the annual research radiation exposure limit.

Ages: 21 Years to 70 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Enrollment: 9 (Actual)
Dates: Start 2005-05; Primary Completion 2007-02 (Actual); Study Completion 2007-02 (Actual)

CONTACTS AND LOCATIONS:
Locations (2):
- United States (2):
  - National Institutes of Health Clinical Center, 9000 Rockville Pike, Bethesda, Maryland
  - Mt. Sinai Medical Center, New York, New York

REFERENCES:
- [Background] Anand A, Charney DS, Oren DA, Berman RM, Hu XS, Cappiello A, Krystal JH. Attenuation of the neuropsychiatric effects of ketamine with lamotrigine: support for hyperglutamatergic effects of N-methyl-D-aspartate receptor antagonists. Arch Gen Psychiatry. 2000 Mar;57(3):270-6. doi: 10.1001/archpsyc.57.3.270. PMID 10711913
- [Background] Austin MP, Mitchell P, Goodwin GM. Cognitive deficits in depression: possible implications for functional neuropathology. Br J Psychiatry. 2001 Mar;178:200-6. doi: 10.1192/bjp.178.3.200. PMID 11230029
- [Background] Austin MP, Mitchell P, Wilhelm K, Parker G, Hickie I, Brodaty H, Chan J, Eyers K, Milic M, Hadzi-Pavlovic D. Cognitive function in depression: a distinct pattern of frontal impairment in melancholia? Psychol Med. 1999 Jan;29(1):73-85. doi: 10.1017/s0033291798007788. PMID 10077295

RESULTS

PARTICIPANT FLOW:
Recruitment Details: Patient with major depression who do not have a serious, unstable medical illness and are 21 to 55 years of age may be eligible. Candidates are screened with a psychiatric and medical history, diagnostic interview, physical examination, electrocardiogram, blood tests and, for women, a pregnancy test.
Pre-assignment Details: Participants are tapered off anti-depression drugs (and any other medications not allowed) over a 3-week period and then begin a 2-week drug-free period. During these 2 weeks they have an electroencephalogram (EEG) with light stimulation, and those whose EEG indicates a seizure disorder are excluded from the study.
Groups:
- Org 24448: Blinded, active experimental compound. Dosing starts at 250 mg once per day for one week, then 250 mg twice per day for one week, then 500 mg twice per day. After 4 weeks with insufficient response, the dose may be increased to 750 mg twice per day. The titration schedule may be delayed if the subject is experiencing adverse effects. The subject may be increased or decreased at the discretion of the investigator. The minimum dose allowed for the study is 250 mg once per day.
- Placebo: Blinded placebo. Dosing starts at 250 mg once per day for one week, then 250 mg twice per day for one week, then 500 mg twice per day. After 4 weeks with insufficient response, the dose may be increased to 750 mg twice per day. The titration schedule may be delayed if the subject is experiencing adverse effects. The subject may be increased or decreased at the discretion of the investigator. The minimum dose allowed for the study is 250 mg once per day.
Period: Overall Study
Arm/Group | Org 24448 | Placebo
Started | 5 | 4
Completed | 2 | 2
Not Completed | 3 | 2

BASELINE CHARACTERISTICS:
Groups:
- Total: Total of all reporting groups
Arm/Group | Org 24448 | Placebo | Total
Number analyzed (Participants) | 5 | 4 | 9
Age, Categorical [Count of Participants; unit: Participants]
  <=18 years | 0 | 0 | 0
  Between 18 and 65 years | 5 | 4 | 9
  >=65 years | 0 | 0 | 0
Age Continuous [Mean (Standard Deviation); unit: years] | 38.20 (7.89) | 40.00 (13.69) | 39.00 (10.11)
Sex: Female, Male [Count of Participants; unit: Participants]
  Female | 3 | 3 | 6
  Male | 2 | 1 | 3
Region of Enrollment [Number; unit: participants]
  United States | 5 | 4 | 9

OUTCOME MEASURES:

1. Primary Outcome: Montgomery-Asberg Depression Rating Scale (MADRS)
Description: The MADRS is a measure of depression severity examined on a weekly basis. The minimum score on the 10 item scale is 0 indicating no depression. The maximum score is 60 indicating a very severe depression. Scores of 18 and above are generally considered to suggest significant levels of depression.
Time Frame: 8 weeks
Measure: Least Squares Mean (Standard Error); unit: Scores on a scale
Arm/Group | Org 24448 | Placebo
Number analyzed (Participants) | 5 | 4
Scores on a scale | 26.425 (10.628) | 24.205 (12.905)
Statistical Analysis 1: Comparison: Org 24448 vs Placebo; Per protocol, a linear mixed model with a first order autoregressive covariance structure was used. Baseline was included as a covariate. Drug and visit were main effects with an interaction between them included; Test type: Superiority or Other; p = .919, Mixed Models Analysis — The test reported here examines the main effect for placebo versus drug; Mean Difference (Final Values) = 2.220, 95% CI 2-sided [-46.565 to 51.006], Standard Error of Mean 18.867 — A positive value indicates greater depression in the active treatment group compared to placebo

ADVERSE EVENTS:
Arm/Group | Org 24448 | Placebo
Serious Adverse Events (participants affected / at risk) | 1/5 | 0/4
Other Adverse Events (participants affected / at risk) | 2/5 | 3/4
SERIOUS ADVERSE EVENTS; cells are participants affected of the arm's N at risk (number of events):
Term (organ system) | Org 24448 (N=5) | Placebo (N=4)
Decreased white blood cell and absolute neutrophils counts (Blood and lymphatic system disorders) | 1 (1) | 0 (0)
OTHER ADVERSE EVENTS (reported when occurring in more than 5% of participants in an arm); cells are participants affected of the arm's N at risk (number of events):
Term (organ system) | Org 24448 (N=5) | Placebo (N=4)
Increased thirst (Gastrointestinal disorders) | 1 (1) | 1 (1)
Memory problems (Nervous system disorders) | 1 (1) | 0 (0)
Headache (General disorders) | 1 (1) | 2 (2)
Pain (General disorders) | 0 (0) | 3 (3)
Dental problems (General disorders) | 0 (0) | 1 (1) — Patient lost tooth
Fatigue (General disorders) | 0 (0) | 1 (1)
Suicidal ideas (Psychiatric disorders) | 0 (0) | 1 (1)
Dizziness (General disorders) | 1 (1) | 0 (0)
Dry mouth (General disorders) | 1 (1) | 0 (0)

CERTAIN AGREEMENTS:
Principal investigators are sponsor employees: Yes; Agreement restricts PI disclosure of results: No